CLINICAL TRIAL: NCT00218062
Title: Pharmacotherapy Dosing Regimen (Cocaine Dependence Population)
Brief Title: Effectiveness of Modafinil and D-amphetamine in Treating Cocaine Dependent Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joy Schmitz, Professor - PSY-Behavioral Sciences, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-09262-12; P50DA009262-12 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Dextroamphetamine; Modafinil; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- D-Amphetamine 60mg + Therapy (Experimental): During the 16 weeks of outpatient treatment, participants took three capsules daily (two in the morning, one in the afternoon). All active and placebo capsules were identical in appearance and each contained 50mg riboflavin for subsequent evaluation of medication compliance. Medication administration was initiated during a 5 day run-up period. d-Amphetamine sustained release (SR) (Dexedrine Spansules) started at 15 mg (day 1-2), increased to 30mg (day3; 15mg, BID), 45mg (day4; 15mg, TID), and 60mg (day5; 15mg bid plus 30mg qd). A 5-day dose reduction schedule occurred at week 17.
  Manual-based, cognitive-behavioral therapy was provided for 1 hour each week by master's-level therapists. The cognitive-behavioral therapy emphasized relapse prevention and coping skills.
  Interventions: Drug: D-Amphetamine 60mg; Behavioral: Therapy
- Modafinil 400mg + Therapy (Experimental): During the 16 weeks of outpatient treatment, participants took three capsules daily (two in the morning, one in the afternoon). All active and placebo capsules were identical in appearance and each contained 50mg riboflavin for subsequent evaluation of medication compliance. Medication administration was initiated during a 5 day run-up period. Modafinil started at 200mg (day1) and increased to 400mg (days2-5). A 5-day dose reduction schedule occurred at week 17.
  Manual-based, cognitive-behavioral therapy was provided for 1 hour each week by master's-level therapists. The cognitive-behavioral therapy emphasized relapse prevention and coping skills.
  Interventions: Drug: Modafinil 400mg; Behavioral: Therapy
- Modafinil 200mg + D-Amphetamine 30mg + Therapy (Experimental): During the 16 weeks of outpatient treatment, participants took three capsules daily (two in the morning, one in the afternoon). All active and placebo capsules were identical in appearance and each contained 50mg riboflavin for subsequent evaluation of medication compliance. Medication administration was initiated during a 5 day run-up period. For the combination condition, dosages of modafinil and d-amphetamine were escalated to one-half of that for the single medication conditions. A 5-day dose reduction schedule occurred at week 17.
  Manual-based, cognitive-behavioral therapy was provided for 1 hour each week by master's-level therapists. The cognitive-behavioral therapy emphasized relapse prevention and coping skills.
  Interventions: Drug: D-Amphetamine 30mg; Drug: Modafinil 200mg; Behavioral: Therapy
- Placebo + Therapy (Placebo Comparator): During the 16 weeks of outpatient treatment, participants took three capsules daily (two in the morning, one in the afternoon). All active and placebo capsules were identical in appearance and each contained 50mg riboflavin for subsequent evaluation of medication compliance.
  Manual-based, cognitive-behavioral therapy was provided for 1 hour each week by master's-level therapists. The cognitive-behavioral therapy emphasized relapse prevention and coping skills.
  Interventions: Behavioral: Therapy; Drug: Placebo

INTERVENTIONS:
Drug: D-Amphetamine 30mg
  Arms: Modafinil 200mg + D-Amphetamine 30mg + Therapy
Drug: D-Amphetamine 60mg
  Arms: D-Amphetamine 60mg + Therapy
Drug: Modafinil 200mg
  Arms: Modafinil 200mg + D-Amphetamine 30mg + Therapy
Drug: Modafinil 400mg
  Arms: Modafinil 400mg + Therapy
Behavioral: Therapy — Manual-based, cognitive-behavioral therapy was provided for 1 hour each week by master's-level therapists. The cognitive-behavioral therapy emphasized relapse prevention and coping skills.
Drug: Placebo
  Arms: Placebo + Therapy

SUMMARY:
Cocaine dependence is a major public health problem; an effective primary treatment for cocaine dependent individuals has yet to be found. The purpose of this study is to examine the effects of d-amphetamine and modafinil, when given alone and in combination, in treating cocaine dependent individuals.

DETAILED DESCRIPTION:
Cocaine is a strong central nervous system stimulant that is widely abused throughout the United Sates. Due to its widespread use, it is important to develop an effective treatment for cocaine dependence. Modafinil is a glutamate-enhancing agent. D-amphetamine is a central nervous system stimulant that is approved to treat individuals with narcolepsy and attention deficit disorder. Both modafinil and d-amphetamine may be effective treatments for cocaine dependence. The purpose of this study is to examine the effectiveness of modafinil and d-amphetamine, alone and in combination, in treating cocaine dependent individuals.

This study will last 16 weeks. Participants will be randomly assigned to one of four groups: 1) 60 mg dose of d-amphetamine; 2) 400 mg dose of modafinil; 3) 30 mg dose of d-amphetamine combined with 200 mg dose of modafinil; and 4) placebo. All participants will receive 200 mg of modafinil over 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Meets Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-IV (SCID) criteria for cocaine abuse or dependence
* In general good health. Individuals who are HIV-positive will not be excluded if in good general health, unless medication interactions exist.

Exclusion Criteria:

* Meets diagnostic criteria for psychiatric disorders, including other forms of drug dependence, other than nicotine
* Current cardiovascular disease, as determined by an electrocardiogram
* On probation or parole if the circumstances do not allow study completion or if ethical constraints of supervision do not allow confidentiality
* Previously received treatment with d-amphetamine, modafinil, or aripiprazole
* Currently receiving prescribed medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2006-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy M. Schmitz, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States

REFERENCES:
- [Result] Schmitz JM, Rathnayaka N, Green CE, Moeller FG, Dougherty AE, Grabowski J. Combination of Modafinil and d-amphetamine for the Treatment of Cocaine Dependence: A Preliminary Investigation. Front Psychiatry. 2012 Aug 30;3:77. doi: 10.3389/fpsyt.2012.00077. eCollection 2012. PMID 22969732

RESULTS

PARTICIPANT FLOW:
Groups:
- Modafinil 400mg + Therapy: During the 16 weeks of outpatient treatment, participants took three capsules daily (two in the morning, one in the afternoon). All active and placebo capsules were identical in appearance and each contained 50mg riboflavin for subsequent evaluation of medication compliance. Medication administration was initiated during a 5 day run-up period. Modafinil started at 200mg (day1) and increased to 400mg (days2-5). A 5-day dose reduction schedule occurred at week 17.
  Manual-based,cognitive-behavioral therapy was provided for 1 hour each week by master's-level therapists. The cognitive-behavioral therapy emphasized relapse prevention and coping skills.
- Modafinil 200mg + D-Amphetamine 30mg + Therapy: During the 16 weeks of outpatient treatment, participants took three capsules daily (two in the morning, one in the afternoon). All active and placebo capsules were identical in appearance and each contained 50mg riboflavin for subsequent evaluation of medication compliance. Medication administration was initiated during a 5 day run-up period. For the combination condition, dosages of modafinil and d-amphetamine were escalated to one-half of that for the single medication conditions. A 5-day dose reduction schedule occurred at week 17.
  Manual-based,cognitive-behavioral therapy was provided for 1 hour each week by master's-level therapists. The cognitive-behavioral therapy emphasized relapse prevention and coping skills.
- Placebo + Therapy: During the 16 weeks of outpatient treatment, participants took three capsules daily (two in the morning, one in the afternoon). All active and placebo capsules were identical in appearance and each contained 50mg riboflavin for subsequent evaluation of medication compliance.
  Manual-based,cognitive-behavioral therapy was provided for 1 hour each week by master's-level therapists. The cognitive-behavioral therapy emphasized relapse prevention and coping skills.
Period: Overall Study
Arm/Group | D-Amphetamine 60mg + Therapy | Modafinil 400mg + Therapy | Modafinil 200mg + D-Amphetamine 30mg + Therapy | Placebo + Therapy
Started | 22 | 20 | 15 | 16
Received First Dose of Study Medication | 16 | 11 | 10 | 12
Completed | 7 | 4 | 3 | 3
Not Completed | 15 | 16 | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- D-Amphetamine 60mg + Therapy: During the 16 weeks of outpatient treatment, participants took three capsules daily (two in the morning, one in the afternoon). All active and placebo capsules were identical in appearance and each contained 50mg riboflavin for subsequent evaluation of medication compliance. Medication administration was initiated during a 5 day run-up period. d-Amphetamine SR (Dexedrine Spansules) started at 15 mg (day 1-2), increased to 30mg (day3; 15mg, BID), 45mg (day4; 15mg, TID), and 60mg (day5; 15mg bid plus 30mg qd). A 5-day dose reduction schedule occurred at week 17.
  Manual-based, cognitive-behavioral therapy was provided for 1 hour each week by master's-level therapists. The cognitive-behavioral therapy emphasized relapse prevention and coping skills.
- Total: Total of all reporting groups
Arm/Group | D-Amphetamine 60mg + Therapy | Modafinil 400mg + Therapy | Modafinil 200mg + D-Amphetamine 30mg + Therapy | Placebo + Therapy | Total
Number analyzed (Participants) | 22 | 20 | 15 | 16 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (6.5) | 42.6 (8.3) | 41.2 (8.5) | 41.9 (9) | 42 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 4 | 2 | 11
  Male | 21 | 16 | 11 | 14 | 62
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 15 | 16 | 73

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use as Assessed by the Treatment Effectiveness Score (TES), Which is the Total Number of Cocaine-negative Urines During Treatment
Time Frame: 16 weeks
Population: All participants who received the first dose of study medication were included in this analysis.
Measure: Mean (Standard Deviation); unit: number of cocaine negative urines
Arm/Group | D-Amphetamine 60mg + Therapy | Modafinil 400mg + Therapy | Modafinil 200mg + D-Amphetamine 30mg + Therapy | Placebo + Therapy
Number analyzed (Participants) | 16 | 11 | 10 | 12
number of cocaine negative urines | 9.25 (13.45) | 6.09 (8.12) | 6 (7.73) | 4.91 (7.56)

2. Primary Outcome: Retention as Indicated by the Number of Participants Who Completed 16 Weeks of Treatment
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | D-Amphetamine 60mg + Therapy | Modafinil 400mg + Therapy | Modafinil 200mg + D-Amphetamine 30mg + Therapy | Placebo + Therapy
Number analyzed (Participants) | 22 | 20 | 15 | 16
participants | 7 | 4 | 3 | 3

3. Primary Outcome: Retention as Indicated by the Number of Participants Who Remained in the Study
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | D-Amphetamine 60mg + Therapy | Modafinil 400mg + Therapy | Modafinil 200mg + D-Amphetamine 30mg + Therapy | Placebo + Therapy
Number analyzed (Participants) | 22 | 20 | 15 | 16
participants | 7 | 4 | 3 | 3

4. Secondary Outcome: Medication Compliance as Indicated by Percentage of Pills Taken According to Self-report
Time Frame: 16 weeks
Measure: Number; unit: percentage of pills taken
Arm/Group | D-Amphetamine 60mg + Therapy | Modafinil 400mg + Therapy | Modafinil 200mg + D-Amphetamine 30mg + Therapy | Placebo + Therapy
Number analyzed (Participants) | 22 | 20 | 15 | 16
percentage of pills taken | 80.2 | 34.5 | 65.8 | 73.2

5. Secondary Outcome: Medication Compliance as Indicated by Percentage of Riboflavin-positive Urine Samples
Time Frame: 16 weeks
Measure: Number; unit: % of riboflavin-positive urine samples
Arm/Group | D-Amphetamine 60mg + Therapy | Modafinil 400mg + Therapy | Modafinil 200mg + D-Amphetamine 30mg + Therapy | Placebo + Therapy
Number analyzed (Participants) | 22 | 20 | 15 | 16
% of riboflavin-positive urine samples | 67.1 | 70 | 76.8 | 66.7

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | D-Amphetamine 60mg + Therapy | Modafinil 400mg + Therapy | Modafinil 200mg + D-Amphetamine 30mg + Therapy | Placebo + Therapy
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 1/22 | 3/20 | 2/15 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-Amphetamine 60mg + Therapy (N=22) | Modafinil 400mg + Therapy (N=20) | Modafinil 200mg + D-Amphetamine 30mg + Therapy (N=15) | Placebo + Therapy (N=16)
Chest pain (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Change in electrocardiogram (EKG) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
High attrition; Pill-taking burden (3 capsules daily) contributed to medication non-compliance; Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes